CLINICAL TRIAL: NCT06102720
Title: Two-center, Prospective, Randomized, Open-label, Controlled Clinical Trial With Endpoint Evaluation
Brief Title: Efficacy of Colchicine in Preventing Recurrent Stroke in the Patients With Acute Atherothrombotic Ischemic Stroke During Hospitalization
Acronym: COLCHIDA
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mikhail Zykov (Other)
Responsible Party: Sponsor-Investigator, Mikhail Zykov, Principal Investigator, Research Institute for Complex Problems of Cardiovascular Diseases, Russia
Organization: Research Institute for Complex Problems of Cardiovascular Diseases, Russia (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: COLCHIDA_1
Record Dates: First submitted 2023-10-22; First posted 2023-10-26 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: Ischemic Stroke
Keywords: ischemic stroke; low-dose colchicine; clopidogrel
MeSH Terms: conditions — Ischemic Stroke | interventions — Colchicine; Clopidogrel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Colchicine Group (Experimental): All patients in this arm will receive colchicine for 14 days in addition to standard medical care without clopidogrel (acetylsalicylic acid, lipid-lowering, antihypertensive, gastroprotective, hypoglycemic drugs if necessary, lifestyle recommendations, early rehabilitation activities).
  Interventions: Drug: Colchicine
- Clopidogrel treatment group (Active Comparator): All patients in this arm will receive standard treatment including clopidogrel.
  Interventions: Drug: Clopidogrel

INTERVENTIONS:
Drug: Colchicine — Oral colchicine will be initiated with a dose of 0.5 mg per day during 14 days. Acetylsalicylic acid was used as an antiplatelet agent (300 mg on days 1 and continuing with 100 mg/day).
  Arms: Colchicine Group
Drug: Clopidogrel — Dual antiplatelet therapy includes ASA (300 mg on days 1 and continuing with 100 mg/day) and clopidogrel (300 mg on days 1 and continuing with 75 mg/day).
  Arms: Clopidogrel treatment group

SUMMARY:
This study is two-center, prospective, randomized, open-label, controlled, investigator-sponsored study that aims to investigate the efficacy of low-dose colchicine in preventing recurrent stroke in the patients with acute atherothrombotic minor-to-moderate ischemic stroke during hospitalization.

DETAILED DESCRIPTION:
This study is two-center, prospective, randomized, open-label, controlled, investigator-sponsored study that aims to investigate the efficacy of low-dose colchicine in preventing recurrent stroke in the patients with acute atherothrombotic minor-to-moderate ischemic stroke during hospitalization. Patients who were eligible to the inclusion criteria and ineligible to the exclusion criteria will be randomly assigned into two groups by a 1:1 ratio. Patients in one arm will receive colchicine initiated with a dose of 0.5 mg per day during on days 1 through 14. Study visits will be performed on the day of randomization and at discharge. The outcomes were stroke, neurological deterioration, сombined endpoint events (stroke, myocardial infarction and death), bleeding during 14 days of follow-up in an intention-to treat analysis.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent form by patient prior to any study-specific procedure.
2. Patient age over 18 years
3. Presence of ipsilateral lesion of the extracranial artery ≥50% according to the European measurement method ECST or its occlusion, as well as stenosis < 50% with signs of morphological instability of the atherosclerotic plaque (ulceration, hemorrhage into the plaque, intimal flotation, mural thrombus, etc.).
4. Minor neurological deficit (NIHSS score ≤5).
5. The duration of development of stroke symptoms before colchicine taken is no more than 48 hours.
6. Confirmation of the presence of a focus of acute ischemia in the brain according to computed tomography or magnetic resonance imaging of the brain.

Exclusion Criteria:

1. The presence of risk factors and conditions that determine a different pathogenetic subtype of ischemic stroke (atrial fibrillation/flutter, ventricular aneurysm, ets.).
2. Hemorrhagic stroke
3. NIHSS score ≤5.
4. Hospitalization of the patient more than 48 hours from the onset of the disease.
5. Severe anemia, thrombocytopenia, leukopenia.
6. Course of an infectious/viral disease.
7. Concomitant treatment with moderate or strong CYP3A4 inhibitors (clarithromycin, erythromycin, telithromycin, other macrolide antibiotics, ketoconazole, itraconazole, voriconazole, ritonavir, atazanavir, indinavir, other HIV protease inhibitors, verapamil or pilitin disulfazole) inhibitors (cyclosporine) at randomization.
8. Concomitant severe degenerative disease of the nervous system.
9. Concomitant inflammatory or autoimmune disease.
10. Dementia, established mental illness.
11. History of malignancy, known hepatitis B or C, or HIV infection.
12. Swallowing impairment interfering with oral administration of the study drug.
13. Pregnancy or breastfeeding. Women of child-bearing potential who are not willing to use a medically accepted method of contraception that is considered reliable in the judgment of the Investigator.
14. Participation in another clinical study with an investigational product at any time during the 30 days prior to randomization
15. Previous enrolment or randomization in the present study.
16. Decrease renal function with creatinine clearance < 30 ml/min.
17. Presence of contraindications to taking colchicine, acetylsalicylic acid and clopidogrel.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-01-12 (Actual); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-02-01 (Estimated)

PRIMARY OUTCOMES:
Any new stroke events | any time within 14 days
  Incidence of any new ischemic stroke.
Neurological deterioration | any time within 14 days
  Neurological deterioration, defined as an increase in The National Institutes of Health Stroke Scale (NIHSS) of 2 or more. The NIHSS provides a quantitative measure of stroke-related neurologic deficit. The higher the score, the more severe the neurological deficit.

SECONDARY OUTCOMES:
New vascular events | any time within 14 days
  Incidence of any new vascular events, including ischemic stroke, myocardial infarction and vascular death
Bleeding event | any time within 14 days
  Bleeding event that is categorised as severe according to GUSTO (Global Utilization Of Streptokinase And Tpa For Occluded Arteries) bleeding criteria.
Positive functional outcome | any time within 14 days
  A positive functional outcome within 14 days is determined if the Modified Rankin Score (mRS) improves to 0-1 and/or Rivermead Mobility Index (RMI) to 14 -15 points and/or Rehabilitation Routing Scale 0 -1 points.
  The mRS is a 6 point disability scale with possible scores ranging from 0 to 5. A separate category of 6 is usually added for patients who expire.
  The RMI includes fifteen mobility items. A maximum score of 15 is possible: higher scores indicate better mobility performance.
  The rehabilitation routing scale is needed by the doctor to understand whether the patient requires rehabilitation. The maximum number of points is 6. The more points the patient scores, the more severe his condition.

CONTACTS AND LOCATIONS:
Locations (2):
- Russia (2):
  - Research Institute for Complex Issues of Cardiovascular Diseas, Kemerovo, Kemerovo Oblast
  - Sochi City Hospital #4, Sochi, Krasnodar Refion

IPD SHARING:
Plan to Share IPD: No